CLINICAL TRIAL: NCT00769067
Title: A Randomized Phase 2 Trial Of Pf-00299804 Versus Erlotinib For The Treatment Of Advanced Non-small Cell Lung Cancer After Failure Of At Least One Prior Chemotherapy Regimen
Brief Title: A Randomized Trial Of PF-00299804 Taken Orally Versus Erlotinib Taken Orally For Treatment Of Advanced Non-Small Cell Lung Cancer That Has Progressed After One Or Two Prior Chemotherapy Regimen
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A7471028; 2008-005235-14 (EudraCT Number)
Record Dates: First submitted 2008-10-07; First posted 2008-10-08 (Estimated); Results first posted 2015-08-21 (Estimated); Last update posted 2015-10-07 (Estimated); Status verified 2015-09

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Lung cancer; advanced; second or third line
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Neoplasm Metastasis | interventions — Erlotinib Hydrochloride; dacomitinib

ARMS (2):
- A (Active Comparator)
  Interventions: Drug: Erlotinib
- B (Experimental)
  Interventions: Drug: PF-00299804

INTERVENTIONS:
Drug: Erlotinib — Continuous oral dosing at 150 mg daily.
  Arms: A
Drug: PF-00299804 — Continuous oral dosing at 45mg daily
  Arms: B

SUMMARY:
This study will compare PF-00299804 given orally on continuous schedule to the approved drug, erlotinib, in patients whose non-small cell lung cancer has progressed after chemotherapy; patients will be randomized to receive one of these drugs, and followed for efficacy and tolerance of each.

ELIGIBILITY:
Inclusion Criteria:

* advanced measurable Non-Small Cell Lung Cancer (NSCLC);
* progressed after 1-2 prior chemotherapy;
* Eastern Cooperative Oncology Group (ECOG) 0-2;
* tissue available for future KRAS/ EGFR testing

Exclusion Criteria:

* prior Epidermal Growth Factor Receptor (EGFR) targeted therapy;
* active or untreated Central Nervous System (CNS) metastases;

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2008-11; Primary Completion 2010-10 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (58):
- United States (25):
  - Northwest Alabama Cancer Center, Muscle Shoals, Alabama
  - Agajanian Institute of Oncology and Hematology, Montebello, California
  - Bridgeport Hospital, Bridgeport, Connecticut
  - Wittingham Cancer Center @ Norwalk Hospital, Norwalk, Connecticut
  - Medical Oncology & Hematology, P.C., Waterbury, Connecticut
  - Winship Cancer Institute at Grady Health Systems, Atlanta, Georgia
  - Winship Cancer Institute, Emory University, Atlanta, Georgia
  - Winship Cancer Institute at Emory University, Atlanta, Georgia
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Augusta Oncology Associates, P.C., Augusta, Georgia
  - Augusta Oncology Associates, PC, Augusta, Georgia
  - John B. Amos Cancer Center, Columbus, Georgia
  - Georgia Cancer Specialists, Decatur, Georgia
  - The Longstreet Cancer Center, Gainesville, Georgia
  - Central Georgia Cancer Care, P.C., Macon, Georgia
  - Northwest Georgia Oncology Center, Marietta, Georgia
  - Central Georgia Cancer Care, P.C., Warner Robins, Georgia
  - Kootenai Cancer Center at Post Falls, Post Falls, Idaho
  - Kootenai Cancer Center, Post Falls, Idaho
  - Midwestern Regional Medical Center, Zion, Illinois
  - Center for Blood and Cancer Disorders, Bethesda, Maryland
  - Associates in Oncology/Hematology, PC, Rockville, Maryland
  - University of Minnesota Cancer Center, Minneapolis, Minnesota
  - The West Clinic, Memphis, Tennessee
  - Oncology/Hematology Associates, Clarksburg, West Virginia
- Australia (4):
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - St. Vincent's Hospital, Fitzroy, Victoria
  - The Andrew Love Cancer Centre,, Geelong, Victoria
  - Border Medical Oncology, Wodonga, Victoria
- Brazil (4):
  - Irmandade da Santa Casa de Misericordia de Porto Alegre (ISCMPA) - Hospital Santa Rita, Porto Alegre, Rio Grande do Sul
  - Hospital Sao Lucas da PUCRS, Porto Alegre, Rio Grande do Sul
  - FUNDACAO PIO XII Hospital de Cancer de Barretos, Barretos, São Paulo
  - Instituto do Câncer do Estado de São Paulo Octavio Frias de Oliveira - ICESP, São Paulo, São Paulo
- Canada (4):
  - BC Cancer Agency - Vancouver Centre, Vancouver, British Columbia
  - Royal Victoria Hospital, Barrie, Ontario
  - RSM Durham Regional Cancer Centre - Lakeridge Health Oshawa, Oshawa, Ontario
  - The Ottawa Hospital Cancer Centre, Ottawa, Ontario
- Hong Kong (2):
  - Department of Clinical Oncology, Shatin, New Territories
  - Department of Clinical Oncology, Tuen Mun Hospital, Tuenmen, New Territories
- Poland (6):
  - Medex spolka cywilna, Chrzanów
  - ¿KardioDent¿, Krakow
  - "Vesalius" Sp. z o.o., Krakow
  - Zaklad Rentgena i USG Wyrobek spolka jawna, Krakow
  - Niepubliczny Zaklad Opieki Zdrowotnej AVI Centrum Medyczne, Warsaw
  - Centrum Onkologii-Instytut im. Marii Sklodowskiej-Curie, Warsaw
- Ponce School of Medicine / CAIMED Center, Ponce, PR, Puerto Rico
- National Cancer Centre, Singapore, Singapore
- South Korea (3):
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University College of Medicine, Yonsei Cancer Center, Seoul
  - SamsungMedicalCenter,SungkyunkwanUnivSchoolofMedicine,Div. of Hematology-Oncology, Dep. of Medicine, Seoul
- Spain (4):
  - Hospital Son Llatzer, Palma de Mallorca, Balearic Islands
  - Hospital Universitari Germans Trias I Pujol, Badalona, Barcelona
  - Hospital Teresa Herrera, A Coruña, La Coruña
  - Hospital de Cruces, Barakaldo, Vizcaya
- Taiwan (2):
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Chest Department, Taipei
- United Kingdom (2):
  - Christie Hospital NHS Foundation Trust, Manchester
  - Churchill Hospital, Oxford

REFERENCES:
- [Derived] Ramalingam SS, O'Byrne K, Boyer M, Mok T, Janne PA, Zhang H, Liang J, Taylor I, Sbar EI, Paz-Ares L. Dacomitinib versus erlotinib in patients with EGFR-mutated advanced nonsmall-cell lung cancer (NSCLC): pooled subset analyses from two randomized trials. Ann Oncol. 2016 Mar;27(3):423-9. doi: 10.1093/annonc/mdv593. Epub 2016 Jan 13. PMID 26768165

RESULTS

PARTICIPANT FLOW:
Groups:
- Erlotinib: Erlotinib 150 milligram (mg) tablet orally once daily continuously in 28-day cycles until unacceptable toxicity, tumor progression or death.
- Dacomitinib: Dacomitinib (PF-00299804) 45 mg tablet orally once daily continuously in 28-day cycles until unacceptable toxicity, tumor progression or death.
Period: Overall Study
Arm/Group | Erlotinib | Dacomitinib
Started | 94 | 94
Treated | 94 | 93 (One participant was not treated: refused treatment for reason other than an adverse event (AE).)
Completed | 0 | 0
Not Completed | 94 | 94
Not completed — Death | 89 | 86
Not completed — Lost to Follow-up | 3 | 1
Not completed — Study terminated by sponsor | 1 | 3
Not completed — Other | 1 | 3
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all randomized participants with study drug assignment designated according to initial randomization, regardless of treatment received.
Groups:
- Total: Total of all reporting groups
Arm/Group | Erlotinib | Dacomitinib | Total
Number analyzed (Participants) | 94 | 94 | 188
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.1 (12.0) | 59.9 (9.5) | 60.0 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 39 | 77
  Male | 56 | 55 | 111

OUTCOME MEASURES:

1. Secondary Outcome: Categorical Summary of Overall Scale Change in European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30)
Description: EORTC QLQ-C30: included global health status/quality of life (QoL), functional (Fn) scales (physical, role, cognitive, emotional, and social), symptom scales (fatigue, pain, nausea/vomiting), and single items (dyspnea, appetite loss, insomnia, constipation, diarrhea, and financial difficulties). Scores were averaged, transformed to 0-100 scale; higher score for Global Qol/Fn scales=better level of QoL/functioning or higher score for symptom scales/items=greater degree of symptoms. Overall scale change is categorized as Improved (if average scales change from baseline: for Global QoL/Fn scales >=10; for symptom scale/item <=-10), Worsened (if average scales change from baseline: for Global QoL/Fn scales <=-10; for symptom scale/item >=10), and Stable (if average scales change from baseline >-10 but <10 for Global QoL/Fn scales and symptom scale/item) and participants in each category are reported.
Time Frame: Baseline up to Cycle 44 (Week 188)
Population: ITT population: all randomized participants with study drug assignment designated according to initial randomization, regardless of treatment received. "N" (number of participants analyzed): participants who completed at least 1 item at baseline. "n": participants evaluable for specified category for each arm, respectively.
Measure: Number; unit: participants
Arm/Group | Erlotinib | Dacomitinib
Number analyzed (Participants) | 88 | 90
participants
  Global QoL: Improved (n= 85, 85) | 14 | 11
  Global QoL: Worsened (n= 85, 85) | 36 | 34
  Global QoL: Stable (n= 85, 85) | 35 | 40
  Physical Functioning: Improved (n= 86, 88) | 12 | 14
  Physical Functioning: Worsened (n= 86, 88) | 25 | 24
  Physical Functioning: Stable (n= 86, 88) | 49 | 50
  Role Functioning: Improved (n= 86, 88) | 18 | 22
  Role Functioning: Worsened (n= 86, 88) | 38 | 31
  Role Functioning: Stable (n= 86, 88) | 30 | 35
  Cognitive Functioning: Improved (n= 86, 85) | 13 | 15
  Cognitive Functioning: Worsened (n= 86, 85) | 21 | 21
  Cognitive Functioning: Stable (n= 86, 85) | 52 | 49
  Emotional Functioning: Improved (n= 86, 85) | 11 | 21
  Emotional Functioning: Worsened (n= 86, 85) | 27 | 26
  Emotional Functioning: Stable (n= 86, 85) | 48 | 38
  Social Functioning: Improved (n= 86, 85) | 24 | 30
  Social Functioning: Worsened (n= 86, 85) | 30 | 19
  Social Functioning: Stable (n= 86, 85) | 32 | 36
  Fatigue: Improved (n= 86, 87) | 18 | 21
  Fatigue: Worsened (n= 86, 87) | 38 | 35
  Fatigue: Stable (n= 86, 87) | 30 | 31
  Pain: Improved (n= 86, 87) | 19 | 19
  Pain: Worsened (n= 86, 87) | 30 | 34
  Pain: Stable (n= 86, 87) | 37 | 34
  Nausea and Vomiting: Improved (n= 86, 87) | 13 | 13
  Nausea and Vomiting: Worsened (n= 86, 87) | 27 | 26
  Nausea and Vomiting: Stable (n= 86, 87) | 46 | 48
  Dyspnea: Improved (n= 86, 88) | 23 | 25
  Dyspnea: Worsened (n= 86, 88) | 26 | 25
  Dyspnea: Stable (n= 86, 88) | 37 | 38
  Loss of Appetite: Improved (n= 85, 87) | 17 | 19
  Loss of Appetite: Worsened (n= 85, 87) | 41 | 43
  Loss of Appetite: Stable (n= 85, 87) | 27 | 25
  Insomnia: Improved (n= 86, 87) | 23 | 22
  Insomnia: Worsened (n= 86, 87) | 32 | 33
  Insomnia: Stable (n= 86, 87) | 31 | 32
  Constipation: Improved (n= 86, 85) | 25 | 32
  Constipation: Worsened (n= 86, 85) | 16 | 13
  Constipation: Stable (n= 86, 85) | 45 | 40
  Diarrhea: Improved (n= 86, 85) | 6 | 4
  Diarrhea: Worsened (n= 86, 85) | 52 | 67
  Diarrhea: Stable (n= 86, 85) | 28 | 14
  Financial Difficulties: Improved (n= 85, 85) | 18 | 17
  Financial Difficulties: Worsened (n= 85, 85) | 21 | 17
  Financial Difficulties: Stable (n= 85, 85) | 46 | 51

2. Secondary Outcome: Categorical Summary of Overall Scale Change in European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire Lung Cancer Module (EORTC QLQ-LC13)
Description: QLQ-LC13 consisted of 13 questions relating to disease symptoms specific to lung cancer and treatment side effects typical of treatment with chemotherapy and radiotherapy. The 13 questions comprised 1 multi-item scale for dyspnea and 10 single-item symptoms and side effects (coughing, hemoptysis, sore mouth, dysphagia, peripheral neuropathy, alopecia, chest pain, arm pain, other pain, and medicine for pain). Scores averaged, transformed to 0-100 scale; higher symptom score = greater degree of symptoms. Overall scale change is categorized as Improved (if average scales change from baseline <=-10), Worsened (if average scales change from baseline >=10), and Stable (if average scales change from baseline >-10 but <10) and participants in each category are reported.
Time Frame: Baseline up to Cycle 44 (Week 188)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Erlotinib | Dacomitinib
Number analyzed (Participants) | 88 | 89
participants
  Dyspnoea: Improved (n= 85, 87) | 18 | 24
  Dyspnoea: Worsened (n= 85, 87) | 29 | 20
  Dyspnoea: Stable (n= 85, 87) | 38 | 43
  Coughing: Improved (n= 85, 87) | 24 | 37
  Coughing: Worsened (n= 85, 87) | 20 | 20
  Coughing: Stable (n= 85, 87) | 41 | 30
  Haemoptysis: Improved (n= 85, 86) | 5 | 8
  Haemoptysis: Worsened (n= 85, 86) | 10 | 10
  Haemoptysis: Stable (n= 85, 86) | 70 | 68
  Sore mouth: Improved (n= 85, 87) | 3 | 5
  Sore mouth: Worsened (n= 85, 87) | 38 | 58
  Sore mouth: Stable (n= 85, 87) | 44 | 24
  Dysphagia: Improved (n= 85, 87) | 7 | 6
  Dysphagia: Worsened (n= 85, 87) | 24 | 35
  Dysphagia: Stable (n= 85, 87) | 54 | 46
  Peripheral: Improved (n= 85, 87) | 22 | 27
  Peripheral: Worsened (n= 85, 87) | 23 | 20
  Peripheral: Stable (n= 85, 87) | 40 | 40
  Alopecia: Improved (n= 84, 87) | 20 | 21
  Alopecia: Worsened (n= 84, 87) | 13 | 21
  Alopecia: Stable (n= 84, 87) | 51 | 45
  Pain in chest: Improved (n= 85, 87) | 26 | 30
  Pain in chest: Worsened (n= 85, 87) | 21 | 13
  Pain in chest: Stable (n= 85, 87) | 38 | 44
  Pain in arm or Shoulder: Improved (n= 85, 87) | 19 | 28
  Pain in arm or Shoulder: Worsened (n= 85, 87) | 27 | 17
  Pain in arm or Shoulder: Stable (n= 85, 87) | 39 | 42
  Pain in other parts: Improved (n= 83, 86) | 26 | 23
  Pain in other parts: Worsened (n= 83, 86) | 27 | 28
  Pain in other parts: Stable (n= 83, 86) | 30 | 35

3. Secondary Outcome: Dermatology Life Quality Index (DLQI)
Description: DLQI: 10-item questionnaire to measure how much the participant's skin problem has impacted their life over the previous week on following 6 domains: symptoms/feelings (2 questions), daily activities (2 questions), leisure (2 questions), work/school (1 question), personal relationships (2 questions), and treatment (1 question). All questions were answered on a 4-point Likert scale ranging from 0 (not at all/not relevant) to 3 (very much/prevented work or studying). The DLQI total evaluable score was calculated by summing the score of each question and ranged from 0 to 30, where higher scores indicated more quality of life impairment.
Time Frame: Cycle (C) 1 Day (D) 1 (baseline), C1D10-14, D1 of subsequent cycles up to C44
Population: ITT population included all randomized participants with study drug assignment designated according to initial randomization, regardless of treatment received. Here "N" (number of participants analyzed) signifies participants evaluable for this measure; "n" signifies participants evaluable for specified category for each arm, respectively.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Erlotinib | Dacomitinib
Number analyzed (Participants) | 87 | 91
units on a scale
  C1D1 (n= 87, 91) | 0.70 (1.97) | 0.88 (2.38)
  C1D10-14 (n=68, 81) | 4.35 (6.25) | 3.06 (4.94)
  C2D1 (n= 80, 82) | 5.16 (6.29) | 3.91 (4.07)
  C3D1 (n= 63, 63) | 4.08 (5.67) | 5.52 (6.65)
  C4D1 (n= 39, 43) | 3.97 (4.59) | 5.95 (6.38)
  C5D1 (n= 25, 38) | 3.56 (3.61) | 5.37 (6.08)
  C6D1 (n= 16, 27) | 4.13 (4.80) | 5.37 (6.67)
  C7D1 (n= 13, 27) | 4.38 (4.07) | 4.93 (6.54)
  C8D1 (n= 11, 24) | 4.64 (3.14) | 5.33 (6.23)
  C9D1 (n= 11, 19) | 3.82 (3.34) | 4.84 (5.76)
  C10D1 (n= 11, 17) | 3.36 (3.04) | 5.88 (7.37)
  C11D1 (n= 10, 15) | 5.60 (5.13) | 6.73 (7.57)
  C12D1 (n= 7, 14) | 6.71 (5.62) | 5.50 (6.99)
  C13D1 (n= 7, 13) | 5.57 (4.08) | 5.08 (7.90)
  C14D1 (n= 6, 12) | 6.00 (3.95) | 6.00 (7.35)
  C15D1 (n= 6, 12) | 4.67 (3.78) | 5.92 (7.40)
  C16D1 (n= 5, 11) | 5.40 (3.91) | 5.36 (8.18)
  C17D1 (n= 4, 11) | 5.00 (4.24) | 5.55 (7.85)
  C18D1 (n= 4, 10) | 3.00 (2.16) | 7.30 (9.08)
  C19D1 (n= 4, 9) | 4.50 (2.38) | 7.22 (7.73)
  C20D1 (n= 2, 10) | 3.50 (3.54) | 6.50 (8.57)
  C21D1 (n= 2, 9) | 3.50 (2.12) | 7.33 (7.76)
  C22D1 (n= 1, 7) | 1.00 (NA) — No measure of dispersion calculated as there is only 1 participant (n=1) | 2.14 (3.67)
  C23D1 (n= 1, 7) | 1.00 (NA) — No measure of dispersion calculated as there is only 1 participant (n=1) | 3.71 (3.99)
  C24D1 (n= 1, 7) | 3.00 (NA) — No measure of dispersion calculated as there is only 1 participant (n=1) | 2.57 (4.08)
  C25D1 (n= 1, 6) | 8.00 (NA) — No measure of dispersion calculated as there is only 1 participant (n=1) | 2.83 (4.45)
  C26D1 (n= 0, 6) | NA (NA) — No measure of dispersion calculated as there are no participants (n=0) | 2.67 (4.13)
  C27D1 (n= 0, 6) | NA (NA) — No measure of dispersion calculated as there are no participants (n=0) | 3.33 (3.98)
  C28D1 (n= 0, 6) | NA (NA) — No measure of dispersion calculated as there are no participants (n=0) | 3.17 (3.82)
  C29D1 (n= 0, 6) | NA (NA) — No measure of dispersion calculated as there are no participants (n=0) | 5.33 (4.59)
  C30D1 (n= 0, 5) | NA (NA) — No measure of dispersion calculated as there are no participants (n=0) | 4.20 (5.12)
  C31D1 (n= 0, 5) | NA (NA) — No measure of dispersion calculated as there are no participants (n=0) | 4.20 (4.97)
  C32D1 (n= 0, 4) | NA (NA) — No measure of dispersion calculated as there are no participants (n=0) | 2.75 (2.50)
  C33D1 (n= 0, 4) | NA (NA) — No measure of dispersion calculated as there are no participants (n=0) | 3.00 (2.94)
  C34D1 (n= 0, 2) | NA (NA) — No measure of dispersion calculated as there are no participants (n=0) | 4.00 (1.41)
  C35D1 (n= 0, 2) | NA (NA) — No measure of dispersion calculated as there are no participants (n=0) | 12.50 (13.44)
  C36D1 (n= 0, 2) | NA (NA) — No measure of dispersion calculated as there are no participants (n=0) | 1.50 (2.12)
  C37D1 (n= 0, 2) | NA (NA) — No measure of dispersion calculated as there are no participants (n=0) | 1.50 (2.12)
  C38D1 (n= 0, 2) | NA (NA) — No measure of dispersion calculated as there are no participants (n=0) | 0.50 (0.71)
  C39D1 (n= 0, 2) | NA (NA) — No measure of dispersion calculated as there are no participants (n=0) | 0.00 (0.00)
  C40D1 (n= 0, 2) | NA (NA) — No measure of dispersion calculated as there are no participants (n=0) | 0.50 (0.71)
  C41D1 (n= 0, 2) | NA (NA) — No measure of dispersion calculated as there are no participants (n=0) | 0.00 (0.00)
  C42D1 (n= 0, 2) | NA (NA) — No measure of dispersion calculated as there are no participants (n=0) | 0.50 (0.71)
  C43D1 (n= 0, 1) | NA (NA) — No measure of dispersion calculated as there are no participants (n=0) | 3.00 (NA) — No measure of dispersion calculated as there are no participants (n=0)
  C44D1 (n= 0, 0) | NA (NA) — No measure of dispersion calculated as there are no participants (n=0) | NA (NA) — No measure of dispersion calculated as there are no participants (n=0)

4. Other Pre Specified Outcome: Number of Participants With Kirsten Rat Sarcoma (KRAS) and Epidermal Growth Factor Receptor (EGFR) Status and EGFR T790M Mutation
Description: Tumor tissue were analyzed at a sponsor-designated laboratory to investigate KRAS and EGFR status (wild type or mutated). Participants who did not provide samples for central laboratory analysis confirmation were classified as "unknown". Additionally blood specimens were analyzed at a sponsor-designated laboratory for T790M mutation in EGFR.
Time Frame: Baseline
Population: ITT population included all randomized participants with study drug assignment designated according to initial randomization, regardless of treatment received. The participants under the category EGFR T790M Mutation are already included in the EGFR Mutant category.
Measure: Number; unit: participants
Arm/Group | Erlotinib | Dacomitinib
Number analyzed (Participants) | 94 | 94
participants
  EGFR Status: Wild Type | 65 | 58
  EGFR Status: Mutant | 11 | 19
  EGFR T790M Mutation | 0 | 2
  EGFR Status: Unknown | 18 | 17
  KRAS Status: Wild Type | 64 | 57
  KRAS Status: Mutant | 14 | 17
  KRAS Status: Unknown | 16 | 20

5. Other Pre Specified Outcome: Soluble Protein Biomarkers Level
Description: Blood specimens were analyzed at a sponsor-designated laboratory for analysis of shed proteins/receptors related to Human Epidermal Growth Factor Receptor (HER) signaling (EGFR, HER-2, Epithelial-cadherin [E-cadherin]). The data collection after C12D1 was not performed, as there were too few participants across both treatment arms after C12D1.
Time Frame: Cycle (C) 1 Day (D) 1 (baseline), D1 of each subsequent cycle up to end of treatment (up to 121 weeks)
Population: Biomarker analysis population: participants who received >=1 dose and had baseline samples submitted as per Institutional Review Board/Independent Ethics Committee approval and participant consent. "N"(number of participants analyzed): participants evaluable for this measure; "n": participants evaluable at each time-point for each arm respectively.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Erlotinib | Dacomitinib
Number analyzed (Participants) | 76 | 73
nanogram per milliliter (ng/mL)
  EGFR, C1D1 (n= 65, 66) | 49.88 (7.513) | 49.44 (9.286)
  EGFR, C2D1 (n= 76, 73) | 48.87 (6.985) | 41.29 (8.132)
  EGFR, C3D1 (n= 43, 53) | 51.28 (6.925) | 42.39 (8.072)
  EGFR, C4D1 (n= 26, 39) | 49.49 (8.41) | 41.9 (8.793)
  EGFR, C5D1 (n= 16, 29) | 48.58 (5.801) | 41.97 (7.974)
  EGFR, C6D1 (n= 15, 27) | 50.32 (7.073) | 42.82 (8.014)
  EGFR, C7D1 (n= 13, 26) | 52.16 (7.449) | 43.16 (9.13)
  EGFR, C8D1 (n= 10, 21) | 54.74 (10.73) | 44.78 (9.673)
  EGFR, C9D1 (n= 8, 17) | 55.38 (12.888) | 47.89 (10.854)
  EGFR, C10D1 (n= 10, 17) | 54.57 (9.244) | 48.12 (13.105)
  EGFR, C11D1 (n= 7, 14) | 59.63 (14.624) | 50.9 (13.667)
  EGFR, C12D1 (n= 6, 13) | 57.65 (11.503) | 52.39 (12.976)
  HER2, C1D1 (n= 65,66) | 10.89 (15.44) | 8.39 (2.05)
  HER2, C2D1 (n= 76,73) | 9.17 (4.946) | 6.42 (2.12)
  HER2, C3D1 (n= 43,53) | 9.26 (6.383) | 6.17 (1.703)
  HER2, C4D1 (n= 26,39) | 9.51 (6.958) | 6.29 (1.716)
  HER2, C5D1 (n= 16,29) | 7.7 (1.79) | 5.96 (1.342)
  HER2, C6D1 (n= 15,27) | 7.45 (2.414) | 6.34 (1.428)
  HER2, C7D1 (n= 13,26) | 8.07 (2.262) | 6.47 (1.773)
  HER2, C8D1 (n= 10,21) | 7.28 (1.279) | 7.15 (3.168)
  HER2, C9D1 (n= 8,17) | 7.32 (1.204) | 6.87 (2.205)
  HER2, C10D1 (n= 10,17) | 7.49 (1.618) | 7.25 (2.883)
  HER2, C11D1 (n= 7,14) | 7.76 (1.735) | 6.56 (1.333)
  HER2, C12D1 (n= 6,13) | 7.15 (1.57) | 6.57 (1.587)
  E-cadherin, C1D1 (n= 65,66) | 51.71 (14.63) | 56.13 (22.694)
  E-cadherin, C2D1 (n= 76,73) | 41.46 (14.982) | 45.4 (18.149)
  E-cadherin, C3D1 (n= 43,53) | 42.58 (13.284) | 42.28 (17.81)
  E-cadherin, C4D1 (n= 26,39) | 40.51 (12.384) | 40.15 (16.105)
  E-cadherin, C5D1 (n= 16,29) | 37.58 (9.951) | 38.15 (10.913)
  E-cadherin, C6D1 (n= 15,27) | 36.78 (7.695) | 39.16 (10.301)
  E-cadherin, C7D1 (n= 13,26) | 38.33 (9.675) | 39.47 (11.977)
  E-cadherin, C8D1 (n= 10,21) | 43.6 (11.661) | 40.94 (13.698)
  E-cadherin, C9D1 (n= 8,17) | 40.26 (8.146) | 38.97 (12.517)
  E-cadherin, C10D1 (n= 10,17) | 40.29 (15.742) | 45.85 (12.244)
  E-cadherin, C11D1 (n= 7,14) | 35.9 (9.239) | 39.44 (8.968)
  E-cadherin, C12D1 (n= 6,13) | 35.48 (8.637) | 40.3 (12.433)

6. Other Pre Specified Outcome: Trough Plasma Concentration (Ctrough) of Dacomitinib (PF-00299804)
Description: Only participants from "Dacomitinib" treatment arm were planned to be analyzed for this outcome.
Time Frame: C1D10-14, C2D1, C3D1, C4D1
Population: Pharmacokinetic (PK) analysis population: all participants who received >=1 dose of study medication, with treatment assignments designated according to actual study treatment received, and from whom at least 1 PK sample was obtained. Here "n" signifies participants who were evaluable at specified time-point.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Dacomitinib
Number analyzed (Participants) | 63
ng/mL
  C1D10-14 (n= 63) | 71.94 (37.496)
  C2D1 (n= 60) | 65.50 (33.292)
  C3D1 (n= 44) | 59.28 (30.089)
  C4D1 (n= 31) | 57.79 (26.206)

7. Primary Outcome: Progression-Free Survival (PFS)
Description: PFS: Time in weeks from randomization to date of objective disease progression or death due to any cause, whichever occurred first. PFS was calculated as (first event date or last known event-free date [if the event date unavailable] minus the date of randomization plus 1) divided by 7. Objective progression is defined using Response Evaluation Criteria in Solid Tumors (RECIST), as at least 20 percent (%) increase in the sum of longest dimensions (LDs) of target lesions, taking as reference the smallest sum of LD recorded since the treatment started and/or unequivocal progression of existing non-target lesions and/or appearance of 1 or more new lesions.
Time Frame: Baseline until disease progression or death, assessed at Cycle 2, 3, 4, 5, 6, thereafter every other cycle up to end of treatment (121 weeks), followed by every 8 weeks >284 weeks
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Erlotinib | Dacomitinib
Number analyzed (Participants) | 94 | 94
weeks | 8.3 [7.9 to 11.7] | 12.4 [8.1 to 16.1]
Statistical Analysis 1: Comparison: Erlotinib vs Dacomitinib; Total 128 events (progression/death) provided 80% power to detect a hazard ratio (HR) of 1.45 (Erlotinib versus Dacomitinib arm) with 1-sided alpha=0.10.This represented a 45% improvement in true median PFS. HR and 95% confidence interval estimated from stratified Cox Regression;2-sided p-value was based on stratified log-rank test with epidermal growth factor receptor (EGFR) status, Kirsten Rat Sarcoma status (KRAS), baseline Eastern Cooperative Oncology Group (ECOG) as stratification factors; Test type: Superiority or Other; p = 0.012, Log Rank — 2-Sided; Adjusted for the stratification factors: EGFR status, KRAS status and baseline ECOG performance status; Hazard Ratio (HR) = 0.657, 95% CI 2-sided [0.472 to 0.914] — The estimated HR was for the Dacomitinib arm versus the Erlotinib arm

8. Secondary Outcome: Percentage of Participants With Objective Response
Description: Percentage of participants with objective response based on assessment of confirmed complete response (CR) or confirmed partial response (PR) according to RECIST version 1.0. CR: disappearance of all target and non-target lesions. PR: at least 30 % decrease in sum of the LDs of target lesion, taking as reference the baseline sum LD. Confirmed responses are those that persist on repeat imaging study at least 4 weeks after initial documentation of response.
Time Frame: as for outcome 7
Population: ITT population included all randomized participants with study drug assignment designated according to initial randomization, regardless of treatment received.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Erlotinib | Dacomitinib
Number analyzed (Participants) | 94 | 94
percentage of participants | 5.3 [1.7 to 12.0] | 17.0 [10.1 to 26.2]
Statistical Analysis 1: Comparison: Erlotinib vs Dacomitinib; Test type: Superiority or Other; p = 0.011, Chi-squared — 2-Sided; Unadjusted

9. Secondary Outcome: Best Overall Response (BOR)
Description: Number of participants with BOR according to RECIST version 1.0: CR= disappearance of all target and non-target lesions. PR= at least 30% decrease in sum of LDs of target lesion, taking as reference baseline sum LD. Stable/no response= neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum of LDs since treatment started. Objective progression= at least a 20% increase in sum of LDs of target lesions, taking as reference the smallest sum of LDs recorded since treatment started and/or unequivocal progression of existing non-target lesions and/or appearance of 1 or more new lesions.
Time Frame: as for outcome 7
Population: as for outcome 8
Measure: Number; unit: participants
Arm/Group | Erlotinib | Dacomitinib
Number analyzed (Participants) | 94 | 94
participants
  Complete Response | 0 | 1
  Partial Response | 5 | 15
  Stable/No Response | 37 | 32
  Objective Progression | 49 | 30
  Indeterminate | 3 | 16

10. Secondary Outcome: Duration of Response (DR)
Description: Time in weeks from first documentation of objective tumor response to objective tumor progression or symptomatic deterioration or death due to any cause, whichever occurred first. Duration of tumor response was calculated as (the date of the first documentation of objective tumor progression or symptomatic deterioration or death due to any cause or last known progression-free date [if none of the event dates available] minus the date of the first CR or PR [which ever occurred first] that was subsequently confirmed plus 1) divided by 7. DR was calculated for the subgroup of participants with a confirmed objective tumor response.
Time Frame: as for outcome 7
Population: Analysis population included sub-set of participants from ITT population who had a confirmed objective tumor response (CR or PR).
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Erlotinib | Dacomitinib
Number analyzed (Participants) | 5 | 16
weeks | 40.1 [24.7 to 72.0] | 71.9 [23.6 to 112.1]

11. Secondary Outcome: Overall Survival (OS)
Description: Time in weeks from randomization to date of death due to any cause. OS was calculated as (the death date or last known alive date (if death date unavailable) minus the date of randomization plus 1) divided by 7.
Time Frame: Baseline until end of treatment (15 August 2014); followed up every 8 weeks after discontinuation from study treatment.
Population: as for outcome 8
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Erlotinib | Dacomitinib
Number analyzed (Participants) | 94 | 94
weeks | 32.3 [24.0 to 40.3] | 41.4 [30.4 to 48.1]
Statistical Analysis 1: Comparison: Erlotinib vs Dacomitinib; HR and its 95% confidence interval were estimated from stratified Cox Regression and 2-sided p-value was based on the stratified log-rank test with EGFR status, KRAS status and baseline ECOG as stratification factors; Test type: Superiority or Other; p = 0.252, Log Rank — 2-Sided; Adjusted by stratification factors: EGFR status, KRAS status and baseline ECOG performance status; Hazard Ratio (HR) = 0.822, 95% CI 2-sided [0.587 to 1.151] — The estimated HR was for the Dacomitinib arm versus the Erlotinib arm

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were recorded from the time that the participant provided informed consent through and including 28 calendar days after the last administration of the investigational product.
Description: The same event may appear as both an AE and a serious AE (SAE). However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Arm/Group | Erlotinib | Dacomitinib
Serious Adverse Events (participants affected / at risk) | 30/94 | 34/93
Other Adverse Events (participants affected / at risk) | 93/94 | 93/93
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib (N=94) | Dacomitinib (N=93)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 2
Chest pain (General disorders) | 1 | 0
Disease progression (General disorders) | 12 | 9
Fatigue (General disorders) | 0 | 1
Malaise (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1
Abscess (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1
Infected dermal cyst (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 0 | 1
Parotitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 4 | 6
Pneumonia bacterial (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Cachexia (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Altered state of consciousness (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 2
Mental status changes (Psychiatric disorders) | 1 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 1
Cyst (General disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 8
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib (N=94) | Dacomitinib (N=93)
Anaemia (Blood and lymphatic system disorders) | 5 | 6
Dry eye (Eye disorders) | 3 | 6
Abdominal pain upper (Gastrointestinal disorders) | 7 | 2
Cheilitis (Gastrointestinal disorders) | 1 | 5
Constipation (Gastrointestinal disorders) | 12 | 9
Diarrhoea (Gastrointestinal disorders) | 46 | 67
Dry mouth (Gastrointestinal disorders) | 8 | 9
Dyspepsia (Gastrointestinal disorders) | 8 | 3
Mouth ulceration (Gastrointestinal disorders) | 5 | 3
Nausea (Gastrointestinal disorders) | 21 | 20
Stomatitis (Gastrointestinal disorders) | 10 | 27
Vomiting (Gastrointestinal disorders) | 14 | 11
Asthenia (General disorders) | 11 | 13
Chest pain (General disorders) | 13 | 5
Fatigue (General disorders) | 33 | 24
Mucosal inflammation (General disorders) | 7 | 23
Oedema peripheral (General disorders) | 4 | 6
Pain (General disorders) | 6 | 5
Conjunctivitis (Eye disorders) | 3 | 9
Paronychia (Infections and infestations) | 8 | 24
Upper respiratory tract infection (Infections and infestations) | 6 | 3
Urinary tract infection (Infections and infestations) | 6 | 5
Weight decreased (Investigations) | 13 | 18
Decreased appetite (Metabolism and nutrition disorders) | 29 | 27
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 11
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 5
Dizziness (Nervous system disorders) | 9 | 3
Dysgeusia (Nervous system disorders) | 7 | 7
Headache (Nervous system disorders) | 8 | 3
Insomnia (Psychiatric disorders) | 5 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 21 | 17
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 16 | 20
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 7
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 | 9
Acne (Skin and subcutaneous tissue disorders) | 11 | 12
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 9
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 54 | 60
Dry skin (Skin and subcutaneous tissue disorders) | 15 | 22
Erythema multiforme (Skin and subcutaneous tissue disorders) | 4 | 10
Exfoliative rash (Skin and subcutaneous tissue disorders) | 14 | 16
Nail disorder (Skin and subcutaneous tissue disorders) | 1 | 7
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 5 | 11
Pruritus (Skin and subcutaneous tissue disorders) | 15 | 14
Skin fissures (Skin and subcutaneous tissue disorders) | 2 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.